CLINICAL TRIAL: NCT03633344
Title: Efficacy of the Administration of Colloidal Silicon Dioxide in Tablet Dosage Form (Carbowhite) in Patients With Acute Diarrhea.
Brief Title: Efficacy of the Administration of Colloidal Silicon Dioxide in Tablet Dosage Form in Patients With Acute Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omnifarma Kiev LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRID CODE-7-180
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2018-08

CONDITIONS: Diarrhoea;Acute
Keywords: Diarrhoea; Carbowhite; Colloidal silicon dioxide
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbowhite (Active Comparator): 3 tablets as a single dose (210 mg х 3 = 630 mg) TID (630 mg х 3 = 1,890 mg)
  Interventions: Drug: Carbowhite
- Carbowhite placebo (Placebo Comparator): 3 tablets as a single dose (210 mg х 3 = 630 mg) TID (630 mg х 3 = 1,890 mg)
  Interventions: Drug: Carbowhite placebo

INTERVENTIONS:
Drug: Carbowhite
  Other Names: Colloidal Silicon Dioxide
  Arms: Carbowhite
Drug: Carbowhite placebo
  Other Names: Placebo
  Arms: Carbowhite placebo

SUMMARY:
The purpose of the study is to demonstrate the antidiarrheal efficacy of colloidal silicon dioxide in tablet dosage form (Carbowhite) in patients with acute diarrhea.

DETAILED DESCRIPTION:
Background: Diarrhea is a medical condition characterized by frequent stool, more than 3 times (and more than 5-7 times in newborns) within the last 24 hours, and/or loose stool. The fecal matter is liquid, its daily mass exceeds 200 g per day, and water content reaches 95%.

Objectives: To demonstrate the antidiarrheal efficacy of colloidal silicon dioxide in tablet dosage form (Carbowhite) in patients with acute diarrhea.

Methods: A randomized clinical trial, double-blind, placebo-controlled, multi-center.

ELIGIBILITY:
Inclusion Criteria:

* signed Informed Consent Form for patient's study participation
* male and female patients at the ages from 18 to 55 years
* acute diarrhea (more than three episodes of liquid stool a day) within 48 hours or less in patients with usually normal stool
* body temperature of ≤ 38 °C
* patient's ability to adequately cooperate in the process of study

Exclusion Criteria:

* aged of <18 or >55 years;
* blood or pus in stool;
* body temperature of >38 °C;
* episodes of acute diarrhea for the last 30 days;
* administration of antidiarrheal products for the last 24 hours;
* salmonellosis (Salmonella of any serotype different from S. typhi and S. paratyphi; ICD-10: A02.0), dysentery (Shigella dysenteriae, Shigella flexneri, Shigella boydii; ICD-10: A03.0-A03.3), colibacillosis (Escherichia coli; ICD-10: A04.0-A04.4) which require administration of antimicrobial products;
* pregnancy, lactation;
* concomitant decompensated diseases or acute conditions which, according to an investigator, may affect study results
* alcoholism and drug abuse;
* participation in any other clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Kurchenko, Study Director — Omnifarma Kyiv LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the study recruited 145 patients. One (1) of the patients dropped out of the study before being randomized.
Groups:
- Carbowhite: 3 tablets as a single dose (210 mg х 3 = 630 mg) TID (630 mg х 3 = 1,890 mg)
  Carbowhite
- Carbowhite Placebo: 3 tablets as a single dose (210 mg х 3 = 630 mg) TID (630 mg х 3 = 1,890 mg)
  Carbowhite placebo
Period: Overall Study
Arm/Group | Carbowhite | Carbowhite Placebo
Started | 120 | 24
Completed | 120 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carbowhite | Carbowhite Placebo | Total
Number analyzed (Participants) | 120 | 24 | 144
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 30.9 [22.9 to 35.0] | 34.8 [23.9 to 47.6] | 31.5 [23.5 to 35.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 12 | 59
  Male | 73 | 12 | 85
Region of Enrollment [Count of Participants; unit: Participants]
  Ukraine | 120 | 24 | 144

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Frequency of Defecation to 3 Times Per Day
Description: Percent of patients administered the investigational production who achieved the efficacy endpoint (reduction in frequency of defecation to 3 times per day, absence of loose stool) on Day 5 or earlier
Time Frame: From randomisation up to 5 days
Measure: Count of Participants; unit: Participants
Groups:
- Carbowhite Placebo: 3 tablets as a single dose (210 mg х 3 = 630 mg) t.i.d. (630 mg х 3 = 1,890 mg)
Arm/Group | Carbowhite | Carbowhite Placebo
Number analyzed (Participants) | 120 | 24
Participants | 118 | 24

2. Secondary Outcome: Compliance Rate
Description: Percent of patients administered the investigational production who discontinued the study
Time Frame: From randomisation up to 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Carbowhite | Carbowhite Placebo
Number analyzed (Participants) | 120 | 24
Participants | 0 | 0

3. Secondary Outcome: Duration of Treatment
Description: Mean duration of treatment
Time Frame: From randomisation up to 5 days
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Carbowhite | Carbowhite Placebo
Number analyzed (Participants) | 120 | 24
days | 1.7 [1.6 to 1.9] | 2.6 [2.3 to 3.0]

4. Secondary Outcome: Quantity of Used Medication
Description: Mean quantity of tablets per treatment course
Time Frame: From randomisation up to 5 days
Measure: Median (Inter-Quartile Range); unit: tablets
Groups:
- Carbowhite Placebo: 3 tablets as a single dose (210mg х 3 = 630 mg) t.i.d. (630 mg х 3 = 1,890 mg);
Arm/Group | Carbowhite | Carbowhite Placebo
Number analyzed (Participants) | 120 | 24
tablets | 12 [12 to 24] | 36 [24 to 48]

ADVERSE EVENTS:
Arm/Group | Carbowhite | Carbowhite Placebo
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/24
Other Adverse Events (participants affected / at risk) | 0/120 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-06-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03633344/Prot_SAP_ICF_000.pdf